CLINICAL TRIAL: NCT02801981
Title: A Double-blind, Randomized, Placebo Controlled, Dose Escalating Crossover Study to Evaluate the Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Parameters of Single Doses of GSK2330672 in Japanese Healthy Male Volunteers
Brief Title: Dose-escalation Study of GSK2330672 in Japanese Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 205808
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Last update posted 2016-11-09 (Estimated); Status verified 2016-11

CONDITIONS: Cholestasis
Keywords: tolerability; healthy volunteers; Cholestasis; safety
MeSH Terms: conditions — Cholestasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Sequence 1: GSK2230672 10mg, 30mg, 90mg, and Placebo (Experimental): Subjects will receive GSK2230672 10 mg in period 1, GSK2230672 30 mg in Period 2, GSK2230672 90 mg in Period 3 and placebo in period 4.
  Interventions: Drug: GSK2230672; Drug: Placebo
- Sequence 2:GSK2230672 10mg, 30mg, Placebo, and GSK2230672 90mg (Experimental): Subjects will receive GSK2230672 10 mg in period 1, GSK2230672 30 mg in Period 2, placebo in period 3, and GSK2230672 90 mg in period 4.
  Interventions: Drug: GSK2230672; Drug: Placebo
- Sequence 3:GSK2230672 10mg, Placebo, GSK2230672 90mg and 180mg (Experimental): Subjects will receive GSK2230672 10 mg in period 1, placebo in Period 2, GSK2230672 90 mg in Period 3 and GSK2230672 180 mg in period 4.
  Interventions: Drug: GSK2230672; Drug: Placebo
- Sequence 4: Placebo, GSK2230672 30mg, 90mg and 180mg (Experimental): Subjects will receive placebo in period 1, GSK2230672 30 mg in Period 2, GSK2230672 90 mg in Period 3 and GSK2230672 180 mg in period 4.
  Interventions: Drug: GSK2230672; Drug: Placebo

INTERVENTIONS:
Drug: GSK2230672 — It will be supplied as white to slightly colored, round, film coated tablet for oral administration containing 10 mg or 45 mg of GSK2330672.
Drug: Placebo — It will be supplied as placebo tablets (with no GSK2230672) visually matching to GSK2230672

SUMMARY:
This study will be the first to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics following single dose of 10 milligrams (mg) to 180 mg of GSK2330672 in Japanese healthy subjects. This is a double-blind, randomized, placebo-controlled, dose-escalating and incomplete block crossover study to be conducted in 16 Japanese healthy subjects. Study will be conducted in four periods; subjects will receive either placebo or GSK2330672 (10 mg, 30 mg, 90 mg or 180 mg based on randomization) in each treatment period. Each period will be separated by washout period (at least 6 days from dosing). Total duration of study for each subject will be approximately 5 weeks from the first dosing to follow up visit.

ELIGIBILITY:
Inclusion Criteria:

* Japanese male aged between 20 and 64 years of age inclusive, at the time of signing the informed consent
* Healthy as determined by the investigator or medically qualified designee based on a medical evaluation including medical history, physical examination, laboratory tests and 12-lead ECG. A subject with a clinical abnormality or laboratory parameter(s) which is/are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the investigator (in consultation with the Medical Monitor if required) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Regular bowel movement >=1 per two days.
* Body weight >= 50 kilogram and body mass index (BMI) is more than or equal to 18.5 kilogram / square meter (kg/m^2) and less than 25.0 kg/m^2
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the consent form and in this protocol.

Exclusion Criteria:

* Alanine transaminase (ALT) and/or bilirubin >1.5x Upper limit of normal (ULN) (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome)
* QT interval corrected for heart rate according to Fridericia's formula (QTcF) > 450 millisecond (msec)
* Current or chronic history of inflammatory bowel disease, chronic diarrhea, Crohn's disease or malabsorption syndromes.
* Current or chronic history of cholelithiasis, inflammatory gall bladder disease, cholestatic liver injury, and cholecystecomy.
* Fecal occult blood test positive at screening.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (includes St. John's Wort) within 14 days or 5 half-lives, whichever is longer, prior to the first dose of study medication.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >14 drinks. One drink is equivalent to 12 grams (g) of alcohol: 350 millilitre (mL) of beer, 150 mL of wine or 45 mL of 80 proof distilled spirits.
* History or regular use of tobacco- or nicotine-containing products within 6 months prior to screening.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation
* A positive pre-study syphilis, Hepatitis B surface antigen, Hepatitis C antibody, Human Immunodeficiency Virus (HIV) antigen antibody or Human T-cell Lymphotropic Virus-1 (HTLV-1) antibody result of screening
* A positive pre-study urine drug screen.
* History of donation of blood or blood products >= 400 mL within 3 months or >= 200 mL within 1 month prior to screening.
* The subject has participated in a clinical trial and has received an investigational product within four months or 5 half-lives (whichever is longer) prior to the dosing day in the current study
* Exposure to more than four new chemical entities within 12 months prior to the dosing day.

Ages: 20 Years to 64 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Number of Subjects with Adverse events (AE) | Maximum of 5 weeks
Safety as assessed by blood pressure | Maximum of 5 weeks
  Systolic and diastolic blood pressure will be measured on Day -1, post dose 2 hours (hrs), 12.5 hrs, 24.5 hrs and at 48 hrs in each period and at follow-up.
Safety as assessed by heart rate | Maximum of 5 weeks
  Heart rate will be measured on Day -1, post dose 2 hrs, 12.5 hrs, 24.5 hrs and at 48 hrs in each period and at follow-up.
Safety as assessed by body temperature | Maximum of 5 weeks
  Body temperature will be measured on Day -1, post dose 2 hrs, 12.5 hrs, 24.5 hrs and at 48 hrs in each period and at follow-up.
Safety as assessed by clinical chemistry parameters | Maximum of 5 weeks
  Blood sample will be collected on Day -1, at 48 hrs in each period and at follow-up
Safety as assessed by haematology | Maximum of 5 weeks
  Blood sample will be collected on Day -1, at 48 hrs in each period and at follow-up
Safety as assessed by urinalysis | Maximum of 5 weeks
  Sample will be collected on Day -1, at 48 hrs in each period and at follow-up
Safety as assessed by fecal occult blood | Maximum of 5 weeks
  Fecal occult blood testing will be conducted on Screening (2 samples during Screening period) and each dosing period (anytime from dosing to next dose).
Safety as assessed by Electrocardiogram (ECG) | Maximum of 5 weeks
  Electrocardiogram will be measured on Day -1, post dose 2 hrs, 12.5 hrs, 24.5 hrs and at 48 hrs in each period and at follow-up.

SECONDARY OUTCOMES:
Plasma concentration of GSK2330672 | Blood samples will be collected predose and post dose at 0.5 hrs, 2 hr, 3.5 hr, 5 hr on Day 1 of each period

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Tokyo, Japan